CLINICAL TRIAL: NCT03768830
Title: Impact of 8-weeks Mild Exercise Training on "Invisible" Symptoms and Quality of Life in Ambulatory and Non-ambulatory (EDSS From 0.0 - 8.0) Individuals With Multiple Sclerosis: a Randomized Controlled Trial
Brief Title: Impact of Exercise on "Invisible" Symptoms and Quality of Life in Multiple Sclerosis Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rijeka (Other)
Responsible Party: Principal Investigator, Tanja Grubic Kezele, Principal Investigator, University of Rijeka
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 003-08/18-01/05
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis; Quality of Life; Motivation; Pain; Headache; Migraine; Anxiety Disorders; Depressive Disorder; Sleep Disorder; Insomnia; Physical Disability; Fatigue
Keywords: Quality of life; Multiple Sclerosis; Pain; Headache; Anxiety Disorders; Depressive Disorder; Sleep Disorder; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Pain; Headache; Migraine Disorders; Anxiety Disorders; Depressive Disorder; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders; Fatigue | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomly selected into 4 groups: MS individuals that will exercise - group (MSE), with related control group of individuals who will not exercise) (MSC).
  In addition, a group of healthy control subjects without MS (HE) will also exercise and be evaluated after the study with related control individuals who will not exercise (HC).
  Group of MS and healthy individuals will exercise under the guidance of a physiotherapist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Multiple Sclerosis Exercise (Experimental): Ambulatory and non-ambulatory MS individuals that will exercise-group (MSE). Intervention is exercise training.
  Interventions: Behavioral: Exercise training
- Multiple Sclerosis Control (no-Exercise) (No Intervention): Ambulatory and non-ambulatory MS individuals that will not exercise-group (MSC).
- Healthy Exercise (Experimental): Healthy individuals that will exercise-group (HE). Intervention is exercise training.
  Interventions: Behavioral: Exercise training
- Healthy Control (no-Exercise) (No Intervention): Healthy individuals that will not exercise (HC).

INTERVENTIONS:
Behavioral: Exercise training — Exercise program includes breathing and upper and lower limbs exercise.
  Arms: Healthy Exercise; Multiple Sclerosis Exercise

SUMMARY:
Patients with multiple sclerosis (MS) struggle on a daily basis with accompanying, "Invisible" symptoms like primary fatigue, pain and emotional-cognitive disorders. With the disease progression, these symptoms only intensify, and in combination with basic physical symptoms, quality of life (QOL) rapidly decreases.

An important goal of researchers and clinicians involves improving the QOL of individuals with MS, and the exercise therapy represents potentially modifiable behavior that positively impacts on pathogenesis of MS and these "Invisible" symptoms, thus improving the QOL.

However, the main barrier for its application is low motivational level that MS patients experience due to fatigue with adjacent reduced exercise tolerability and mobility, and muscle weakness. Getting individuals with MS motivated to engage in continuous physical activity may be particularly difficult and challenging, especially those with severe disability or Expanded Disability Status Scale (EDSS 6-8).

Till now, researchers have focused their attention mainly on the moderate or vigorous intensity of exercise and on cardiorespiratory training in MS patients to achieve improvements in daily life quality, less indicating the exercise content, and most importantly, breathing exercises.

In addition, it is investigators intention to make exercise for MS patients more applicable and accessible, motivational and easier, but most important, productive.

Investigators think that MS patients experience more stress with aerobic exercise or moderate to high intensity program exercise, and can hardly keep continuum including endurance exercise, or treadmill.

Hypothesis:

Investigators hypothesis is that 8-weeks of continuous low demanding or mild exercise program with the accent on breathing exercise can attenuate primary fatigue, pain, headaches, emotional-cognitive and sleep dysfunctions in MS patients and provide maintenance of exercise motivation. Investigators also propose that important assistant factor for final goal achievement is social and mental support of the exercise group (EDSS from 0-8) led by a physiotherapist. This will help to maintain exercise motivation and finally make better psychophysical functioning, and thus better QOL.

DETAILED DESCRIPTION:
This study will include individuals with multiple sclerosis including all MS types with EDSS from 0-8, who will be practicing at the Multiple Sclerosis Association in Rijeka for a period of 2 month, 2 times a week for 60 minutes per exercise (total 16h).

Participants will be randomly selected into 2 groups: MS individuals that will exercise - group (MSE), with related control group of individuals who will not exercise) (MSC).

In addition, a group of healthy control subjects without MS (HCE) will also exercise and be evaluated after the study with related control individuals who will not exercise (HCC).

Group of MS and healthy individuals will exercise under the guidance of a physiotherapist. Exercise will be carried out sitting on the chairs for all participants, regardless of whether participants are able to walk or not. The physiotherapist will first demonstrate and explain each exercise. Participants will be emphasized during exercise to stop exercising if there is tiredness, weakness, pain or any other discomfort.

At the beginning of each exercise session, exercise will be initiated by warming muscles and breathing exercises. Therapeutic and abdominal breathing exercises with extended exhalation will be also conducted. Then follow the exercises of stretching and increasing the movement range of the upper and lower limbs. Participants will work with dumbbells and elastic straps to strengthen the muscles of the extremities. In the end of training session, there will be devoted to stretching of the muscle groups involved during exercise.

Each participant involved in the study will undergo the examination through several functional tests at the beginning and up to 8-weeks of the study or exercise, including post-exercise questionnaire for motivation analysis:

1. Assessment of pain level using a "Visual Analogue Scale" for pain (VAS). It is a psychometric response scale or a measurement instrument for subjective characteristics that cannot be directly measured. Here, the participants state their degree of agreement with the facial expression shown with the description of the pain in words, including the appropriate number below the image. The VAS for pain is 5 units long, 0 to 5 (0-no pain and 5-hardest possible pain). Since every patient experiences a pain differently, this simple test can evaluate and make it visible.
2. Assessment of Headache-Migraine intensity and frequency using Headache-Migraine survey.
3. Evaluation of Quality of Life using the abbreviated version of the "36-Item Short Form Survey" (36-SF). It contains 36 questions including 8 subclasses: physical function, role of constraints due to physical problems, physical pain, general health perception, energy level, social function, the role of limitations due to psychological problems and general mental health. The test time is 10 minutes. The scoring system for the SF-36 is relatively complex and is obtained by summing the results for each sub-base separately. Two summaries can be derived from physical subclasses and psychic subclasses. SF-36 is one of "Multiple Sclerosis Quality of Life Inventory" (MSQLI) and Multiple Sclerosis Quality of Life-54(MSQOL-54) .
4. Assessment of psychological distress using the "Clinical Outcomes in Routine Evaluation - Outcome Measure" (CORE-OM). The CORE-OM has 34 items, all with the same five level response choice, and covers the last seven days. It was designed, and this was led partly by the commissioning specification, to cover four main domains: wellbeing, problems, functioning and risk and has 4, 12, 12 and 6 items focused on those domains respectively. The original scoring was the mean across the items, i.e. between 0 and 4 as the scoring of the item responses is from 0 to 4, more recently, to require fewer decimal places, scores have often been reported after multiplying that by ten.
5. Fatigue estimation using the "Modified Fatigue Impact Scale" (MFIS). It is a modified form of the Fatigue Impact Scale based on data obtained from interviews with MS patients on how tiredness affects their lives. This test gives an assessment of tiredness effects on physical, cognitive and psychosocial functioning and can therefore be treated as 3 separate categories. In full-time MFIS consists of 21 questions. The time to complete is 5-10 minutes and the examinee can solve the test without the help of an interviewer. The total points are obtained by summing all the answers or the additions are made separately by the mentioned categories.
6. Assessment the quality of sleep using the Pittsburgh Sleep Quality Index (PSQI). The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month.
7. Assessment the insomnia using the Insomnia Severity Index (ISI). The test is designed to assess the nature, severity, and impact of insomnia and it consists of 7 items: Severity of sleep onset, sleep maintenance and early morning wakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, notice ability of sleep problems by others, distress caused by the sleep difficulties.
8. Questionnaire upon completion of exercise. The final questionnaire will analyze whether the participants really felt health change after exercise cycle and motivated them in a group under the guidance of a physiotherapist to continue self-exercising at home.

Each participant will be familiar with the research protocol to be implemented in accordance with the Code of Ethics and respecting the principles of the Patient Rights. The investigator will explain the use of the tests. Participants will confirm their participation by signing their consent. Participants voluntarily involved in this research will be provided oral and written consent with the explanation of the possibility of giving up at any time during this study without consequences for their further treatment, guaranteed discretion and anonymity of the obtained data.

Statistical data processing:

The results of the research will be statistically analyzed using a computer program of Version 13 (Sigma Plot Scientific Graphing System, v13.0). Statistical significance will be calculated by non-parametric test for dependent samples and parametric test for dependent samples in cases of normal data distribution. Data will be expressed as mean value ± standard error or as a central value of the median value range. The correlation of the observed changes will be investigated by Pearson's correlation for parametric or by Spearman's for non-parametric data. Significant statistical changes will be considered at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with multiple sclerosis (EDSS 0-8)
* Ambulatory and non-ambulatory (in wheelchairs)

Exclusion Criteria:

* Individuals with contraindications for exercising
* Individuals with multiple sclerosis with EDSS over 8

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
Change of fatigue intensity | baseline, up to 8 weeks
  Fatigue estimation using the "Modified Fatigue Impact Scale" (MFIS) questionnaire. This test gives an assessment of tiredness effects on physical, cognitive and psychosocial functioning and can therefore be treated as 3 separate categories. In full-time MFIS consists of 21 questions. The time to complete is 5-10 minutes and the examinee can solve the test without the help of an interviewer. The total points are obtained by summing all the answers or the additions are made separately by the mentioned categories.
Change of pain intensity | baseline, up to 8 weeks
  Assessment of pain level using a "Visual Analogue Scale" (VAS) for pain. It is a psychometric response scale or a measurement instrument for subjective characteristics that cannot be directly measured. Here, the participants state their degree of agreement with the facial expression shown with the description of the pain in words, including the appropriate number below the image. The VAS for pain is 5 units long, 0 to 5 (0-no pain and 5-hardest possible pain).
Change in quality of life | baseline, up to 8 weeks
  Evaluation of Quality of Life using the abbreviated version of the "36-Item Short Form Survey" (36-SF) including physical function, role of constraints due to physical problems, physical pain, general health perception, energy level, social function, the role of limitations due to psychological problems and general mental health.
Change in sleeping quality - ISI | baseline, up to 8 weeks
  Evaluation of sleeping quality using ISI questionnaire. The test is designed to assess the nature, severity, and impact of insomnia and it consists of 7 items: Severity of sleep onset, sleep maintenance and early morning wakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, notice ability of sleep problems by others, distress caused by the sleep difficulties.
Change in sleeping quality - PSQI | baseline, up to 8 weeks
  Evaluation of sleeping quality using PSQI questionnaire. The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring 7 areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month.
Change in psychological symptoms | baseline, up to 8 weeks
  The CORE-OM has 34 items, all with the same five level response choice, and covers the last seven days. It was designed, and this was led partly by the commissioning specification, to cover four main domains: wellbeing, problems, functioning and risk and has 4, 12, 12 and 6 items focused on those domains respectively. The original scoring was the mean across the items, i.e. between 0 and 4 as the scoring of the item responses is from 0 to 4, more recently, to require fewer decimal places, scores have often been reported after multiplying that by ten. Caution should be used to make sure whether results are reported with that x10 multiplier though it is rarely likely that results can be confused as to scoring.
Change in Headache-Migraine intensity and frequency | baseline, up to 8 weeks
  Survey Survey made from questions for subjective self-evaluation of Headache-Migraine intensity and frequency.

SECONDARY OUTCOMES:
Motivation evaluation | up 8 weeks
  Survey made from questions for subjective self-evaluation of motivation efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Grubić Kezele, PhD, MD, Principal Investigator — University of Rijeka
Locations (1):
- University of Rijeka, Faculty of Medicine, Department of Physiology, Immunology and Pathophysiology, Rijeka, Croatia

REFERENCES:
- [Derived] Grubic Kezele T, Trope Z, Ahel V, Ruzic N, Omrcen H, Dudaric L, Fuzinac-Smojver A. Upper-lower limb and breathing exercise program for improving sleep quality and psychological status in multiple sclerosis: a pilot randomized controlled trial. Brain Impair. 2023 Mar;24(1):86-102. doi: 10.1017/BrImp.2021.17. Epub 2021 Oct 1. PMID 38167585